CLINICAL TRIAL: NCT06633692
Title: Female Pelvic Blood Flow Under Simulated Microgravity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceren UNAL (Other)
Responsible Party: Sponsor-Investigator, Ceren UNAL, M.D., Koc University Hospital
Organization: Koc University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024.238.IRB1.028
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Uterine; Ovary; Microgravity; Blood Flow
Keywords: microgravity; female pelvic blood flow; doppler ultrasound
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Intervention Model Description: Pre- and post-assessment of the pelvic blood flow in response to simulated microgravity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulated microgravity (Experimental): Pre- and post-assessment of pelvic blood flow in response to simulated microgravity will be performed in the same participant.
  Interventions: Other: Head down tilt (HDT)

INTERVENTIONS:
Other: Head down tilt (HDT) — In the head-down tilt intervention, a participant is positioned on a tilt table, initially in supine position and afterwards with their head inclined downward at a specific angle. This position causes a shift of body fluids towards the head, mimicking the fluid redistribution observed in microgravity conditions in space.

SUMMARY:
Spaceflight is characterized by unique physiological adaptations. Cardiovascular system response to the microgravity includes major changes. During spaceflight, body fluids are displaced in the cephalad direction due to changes in gravity, resulting in altered vascular dynamics and the redistribution of the blood circulation.

As the investigators approach crewed Moon and Mars missions and commercial spaceflights become more frequent, understanding the impact of space travel on women's health is crucial. Despite the known importance of these vascular dynamics in both clinical and research settings, there is limited information on the pelvic blood flow under microgravity. The aim of this project is to fill this gap by analyzing the impact of simulated microgravity on the perfusion of female reproductive organs using Doppler velocimetry. Head-down tilt (HDT) position is an established model in literature for simulated microgravity on Earth.

This prospective study will assess pelvic organ blood flow in the supine position after a period of acclimation as a control. After completing Doppler measurements in the supine position, the participant will be placed in the HDT position. Following a period of acclimation, Doppler measurements will be repeated on the same vessels.During both supine and simulated microgravity conditions, vital signs (i.e., blood pressure, heart rate, oxygen saturation) will be collected.

DETAILED DESCRIPTION:
Cardiovascular system response to the microgravity includes major changes. During spaceflight, body fluids are displaced in the cephalad direction due to changes in gravity, resulting in altered vascular dynamics and the redistribution of the blood circulation. Redistribution of fluids triggers baroreceptor reflex and autonomic response initiates. Cardiovascular response to the microgravity environment is affected by gender. Women tend to lose more plasma volume and have less peripheral vascular resistance in response to microgravity analogue situations like bed rest.

Simulated microgravity leads to increased stiffness and remodeling of the aorta, a major vessel supplying blood to the abdomen, pelvis, and lower extremities. Pelvic organs are located in the lower abdomen and have rich blood supply through these major blood vessels and anastomosis. Mathematical modeling for microgravity showed a 6% mean flow rate variation in the last part of abdominal aorta. Furthermore, mean flow rate variations and resistance changed based on the branching arteries, such as internal iliac arteries. The uterine and ovarian arteries branch from the internal iliac arteries and abdominal aorta, respectively. Blood supply to an organ and tissue perfusion are vital for the proper functioning of the organs and tissues.

As the investigators approach crewed Moon and Mars missions and commercial spaceflights become more frequent, understanding the impact of space travel on women's health is crucial. Despite the known importance of these vascular dynamics in both clinical and research settings, there is limited information on the pelvic blood flow under microgravity. Our aim is to fill this gap by analyzing the impact of simulated microgravity on the perfusion of female reproductive organs using Doppler velocimetry. Head-down tilt (HDT) position is an established model in literature for simulated microgravity on Earth.

This prospective study will be conducted at Koç University Hospital. Adult women of reproductive age (18-44 years) undergoing abdominal ultrasound will be recruited. Participants will be selected from a cohort presenting for their well-woman visit; there will be no additional visits. Ultrasound and Doppler spectrometry evaluations will be carried out with convex and linear probes of the GE Loqic S8 device. The researchers will assess pelvic organ blood flow in the supine position after a period of acclimation as a control. After completing Doppler measurements in the supine position, the participant will be placed in the HDT position. Following a period of acclimation, Doppler measurements will be repeated on the same vessels. During both supine and simulated microgravity conditions, vital signs (i.e., blood pressure, heart rate, oxygen saturation) will be collected. Pre- and post-HDT Doppler measurements will be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18-44 years old healthy female individuals

Exclusion Criteria:

* History of hysterectomy and/or oophorectomy
* Pregnancy
* Premature ovarian insufficiency
* Women with reproductive tract pathologies
* Cardiovascular diseases

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Internal iliac artery Doppler indices before and after HDT | through study completion, an average of 1 year
  Internal iliac artery Doppler flow indices will be obtained in supine and HDT positions after acclimation periods

SECONDARY OUTCOMES:
Ovarian artery Doppler indices before and after HDT | through study completion, an average of 1 year
  Ovarian artery Doppler flow indices will be obtained in supine and HDT positions after acclimation periods

CONTACTS AND LOCATIONS:
Overall Officials: Afak Durur Karakaya, M.D., Principal Investigator — Koç University
Locations (1):
- Koc Universoty Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Perhonen MA, Franco F, Lane LD, Buckey JC, Blomqvist CG, Zerwekh JE, Peshock RM, Weatherall PT, Levine BD. Cardiac atrophy after bed rest and spaceflight. J Appl Physiol (1985). 2001 Aug;91(2):645-53. doi: 10.1152/jappl.2001.91.2.645. PMID 11457776
- [Background] Waters WW, Ziegler MG, Meck JV. Postspaceflight orthostatic hypotension occurs mostly in women and is predicted by low vascular resistance. J Appl Physiol (1985). 2002 Feb;92(2):586-94. doi: 10.1152/japplphysiol.00544.2001. PMID 11796668
- [Background] Herault S, Fomina G, Alferova I, Kotovskaya A, Poliakov V, Arbeille P. Cardiac, arterial and venous adaptation to weightlessness during 6-month MIR spaceflights with and without thigh cuffs (bracelets). Eur J Appl Physiol. 2000 Mar;81(5):384-90. doi: 10.1007/s004210050058. PMID 10751099
- [Background] Shen M, Frishman WH. Effects of Spaceflight on Cardiovascular Physiology and Health. Cardiol Rev. 2019 May/Jun;27(3):122-126. doi: 10.1097/CRD.0000000000000236. PMID 30365406
- [Background] Gallo C, Ridolfi L, Scarsoglio S. Cardiovascular deconditioning during long-term spaceflight through multiscale modeling. NPJ Microgravity. 2020 Oct 1;6:27. doi: 10.1038/s41526-020-00117-5. eCollection 2020. PMID 33083524
- [Background] Tuday EC, Meck JV, Nyhan D, Shoukas AA, Berkowitz DE. Microgravity-induced changes in aortic stiffness and their role in orthostatic intolerance. J Appl Physiol (1985). 2007 Mar;102(3):853-8. doi: 10.1152/japplphysiol.00950.2006. Epub 2006 Nov 2. PMID 17082368
- [Background] Mathyk B, Imudia A, Quaas A, Halicigil C, Karouia F, Avci P, Nelson N, Guzeloglu-Kayisli O, Denbo M, Sanders L, Scott R, Basar M, Guevara-Cerdan A, Strug M, Monseur B, Kayisli U, Szewczyk N, Mason CE, Young SL, Tasoglu S, Costes S, Beheshti A.Understanding how space travel affects the female reproductive system to the Moon and beyond. npj Womens Health 2, 20 (2024). https://doi.org/10.1038/s44294-024-00009-z